CLINICAL TRIAL: NCT06710613
Title: Efficacy of High-flow Nasal Oxygen in Preventing Hypoxia During Gastrointestinal Endoscopy: a Retrospective Cohort Study
Status: Active, not recruiting | Type: Observational
Sponsor: Fengli Liu (Other)
Responsible Party: Sponsor-Investigator, Fengli Liu, Student, Nanchang University
Organization: Nanchang University (Other)
Other Study IDs: LY2024-275-B
Record Dates: First submitted 2024-11-23; First posted 2024-11-29 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Hypoxia
Keywords: High flow nasal cannula oxygen
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Medical record
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- control group: conventional nasal cannula oxygen group
- experimental group: high flow nasal cannula oxygen group

SUMMARY:
During painless gastroscopy, the occurrence of hypoxia is a critical concern, especially under intravenous anesthesia using propofol. This study aimed to investigate the incidence of hypoxia during painless gastroscopy and evaluate preventive measures.

DETAILED DESCRIPTION:
From June 15 th 2023 to August 15th 2023, 900 patients who underwent elective gastroscopy in the Renji Hospital, Shanghai Jiao Tong University School of Medicine were selected. They were divided into the high flow nasal cannula oxygen group and the conventional nasal cannula oxygen group by oxygen inhalation. Patient demographics, Mallampati class, and other relevant factors were compared between the two groups. Primary outcomes included the incidence hypoxia (SpO2 < 90%), while secondary outcomes included subclinical respiratory depression, and adverse events related to nasal oxygen cannula.

ELIGIBILITY:
Inclusion Criteria：

* Patients aged 18 to 70
* Undergoing painless gastroscopy under intravenous anesthesia

Exclusion Criteria：

* Severe respiratory disease
* History of nasal bleeding or mucosal injury
* Emergency cases
* Pregnant or lactating female

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who underwent painless gastroscopy
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
incidence of hypoxia | 60 seconds
  SpO2 levels less than 90%

SECONDARY OUTCOMES:
the incidence of subclinical respiratory depression and adverse events | 30 minute
  the incidence of and subclinical respiratory depression (SpO2 levels between 90% and less than 95%) and adverse events(mouth or nasal dryness, headache, nasal mucosal injury with bleeding, barotrauma. )

CONTACTS AND LOCATIONS:
Overall Officials: Fengli Liu, master, Principal Investigator — Nanchang University
Locations (1):
- Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No